CLINICAL TRIAL: NCT02555228
Title: Benefits of Premedication With Small Volume Simethicone Solution Before Diagnostic Gastroscopy: A Randomized Endoscopist-blinded Prospective Study
Brief Title: Small Volume Simethicone Before Gastroscopy: Any Benefit?
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Changi General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: CGH-QIPSMJ
Record Dates: First submitted 2015-09-13; First posted 2015-09-21 (Estimated); Results first posted 2016-03-15 (Estimated); Last update posted 2016-03-15 (Estimated); Status verified 2016-02

CONDITIONS: Lesion of Stomach
Keywords: simethicone; gastroscopy; McNalley score
MeSH Terms: interventions — Simethicone; Water

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Simethicone premedication (Experimental): Liquid simethicone (1ml volume) in 5mls of water
  Interventions: Drug: Simethicone
- Placebo (Placebo Comparator): Just 5 mls of water
  Interventions: Other: Water

INTERVENTIONS:
Drug: Simethicone — 100mg of liquid simethicone is put into 5mls of water and given at least 30 minutes before the gastroscopy.
  Arms: Simethicone premedication
Other: Water — 5mls of water is given at least 30 minutes before the gastroscopy.
  Arms: Placebo

SUMMARY:
A randomized controlled and endoscopist-blinded study which compares the efficacy of liquid simethicone (100mg) in 5 mls water, versus placebo ( 5mls of water), as premedication (given at least 30 minutes) before gastroscopy towards improvement of the total mucosal visibility score.

DETAILED DESCRIPTION:
Excessive bubbles or foam during gastroscopy is a common problem which can cause significant hindrance to an optimal evaluation of the gastric mucosa, prolong the procedure time, and contribute to poor patient tolerance during the scope.

Simethicone, with or without N-acetylcysteine, has been extensively evaluated to improve mucosal visibility. However, the volume of simethicone preparation and the timing of ingesting this solution before gastroscope varied significantly across different studies. In general, it appeared that a larger volume of simethicone solution, given earlier before the gastroscopy, may yield better results. However, allowing a patient to ingest a large volume of liquid before a gastroscopy under sedation brings forth the risk of aspiration. A recent Taiwanese study published in 2014 [1] showed that the subgroup with 100mg of simethicone in just 5ml of water, did achieve a good total mucosal visibility score, if the solution was ingested more than 30 minutes before the gastroscope. This may be because a longer time allows the simethicone to coat more of the mucosa. However, this study did not compare this preparation against a placebo.

In Changi General Hospital, many gastroscopies are done daily with no premedication. Also, there is no protocol for premedication before gastroscopes. This study hopes to prove that a low volume of simethicone solution, given at an ample time (more than 30 minutes) before the scope, can significantly improve overall endoscopy performance compared to no premedication at all.

ELIGIBILITY:
Inclusion Criteria:

* Planned for an elective diagnostic gastroscopy by the attending gastroenterologist
* Age of at least 21 years old
* Mentally competent and able to provide informed consent

Exclusion Criteria:

* Category A patients (incarcerated prisoners)
* adults who are unable to give their own informed consent due to lack of mental capacity
* suspected gastrointestinal bleeding
* suspected impacted foreign material
* suspected gastric outlet obstruction
* suspected esophageal obstruction
* history of dysphagia
* known hypersensitivity to simethicone
* previous gastrectomy

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2015-08; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Changi General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Yes
Data send to Singapore Health Sciences Authority

RESULTS

PARTICIPANT FLOW:
Groups:
- Simethicone Premedication: Liquid simethicone (1ml volume) in 5mls of water
  Simethicone: 100mg of liquid simethicone is put into 5mls of water and given at least 30 minutes before the gastroscopy.
  27 patients randomized to this group.
- Placebo: Just 5 mls of water
  Water: 5mls of water is given at least 30 minutes before the gastroscopy.
  27 patients randomized to this group.
Period: Overall Study
Arm/Group | Simethicone Premedication | Placebo
Started | 27 (20th August 2015) | 27 (14th August 2015)
Completed | 27 (19th November 2015) | 27 (29th October 2015)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Simethicone Premedication | Placebo | Total
Number analyzed (Participants) | 27 | 27 | 54
Age, Customized [Mean (Standard Deviation); unit: years]
  Age | 57.7 (12.5) | 52.9 (15.5) | 55.3 (14)
Sex/Gender, Customized [Number; unit: participants]
  Male patients | 15 | 9 | 24
  Female patients | 12 | 18 | 30
Region of Enrollment [Number; unit: participants]
  Singapore | 27 | 27 | 54
Mean premedication time (min:sec) [Mean (Standard Deviation); unit: seconds] | 2686 (756) | 2468 (596) | 2577 (676)

OUTCOME MEASURES:

1. Primary Outcome: Total Cumulative Mucosal Visibility Score
Description: Total cumulative mucosal visibility score (TMVS) of all areas during the gastroscopy as determined by Mc Nally score:
  Score of 1: no bubbles Score of 2: minimal-occasional bubbles; must actively look for them Score of 3: moderate-obviously present Score of 4: severe-so many bubbles that vision is obscured
  Total areas covered:
  (E) esophagus (D) duodenum (A) Antrum and angularis (B) body and fundus
Time Frame: This will be calculated during the diagnostic gastroscopy, an expected duration of 10 minutes.
Measure: Mean (Standard Deviation); unit: units
Arm/Group | Simethicone Premedication | Placebo
Number analyzed (Participants) | 27 | 27
units | 5.78 (1.65) | 8.89 (1.97)

2. Secondary Outcome: Mucosal Visibility Score Per Area as Determined by Mc Nally Score:
Description: * Area E: esophagus
  * Area D: duodenum
  * Area A: antrum and angularis
  * Area B: body and fundus
  Mc Nally score per area:
  Score of 1: no bubbles Score of 2: minimal-occasional bubbles; must actively look for them Score of 3: moderate-obviously present Score of 4: severe-so many bubbles that vision is obscured
Time Frame: This will be calculated during the diagnostic gastroscopy, an expected duration of 10 minutes.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Simethicone Premedication | Placebo
Number analyzed (Participants) | 27 | 27
units on a scale
  Area E (esopahgus) | 1.48 (0.57) | 1.59 (0.57)
  Area D (duodenum) | 1.26 (0.53) | 2.26 (0.81)
  Area A (antrum and angularis) | 1.30 (0.54) | 2.56 (1.05)
  Area B (body and fundus) | 1.74 (0.81) | 2.44 (0.97)

3. Secondary Outcome: Volume of Additional Manual Flushes Required During Endoscopy in Mls
Description: The volume of additional water (in mls) flushed during the gastroscopy in order to remove obscuring foam or bubbles.
Time Frame: This will be calculated during the diagnostic gastroscopy, an expected duration of 10 minutes.
Measure: Mean (Standard Deviation); unit: mls
Arm/Group | Simethicone Premedication | Placebo
Number analyzed (Participants) | 27 | 27
mls | 3.89 (11.46) | 84.81 (110.18)

4. Secondary Outcome: Adverse Events in Each Group Which May or May Not be Related to Simethicone Solution
Time Frame: Participants will be followed from ingestion of the premedication to the time of discharge from the endoscopy center, an estimated duration. of 3 hours
Measure: Number; unit: number of events
Arm/Group | Simethicone Premedication | Placebo
Number analyzed (Participants) | 27 | 27
number of events | 0 | 0

ADVERSE EVENTS:
Time Frame: Any adverse event that occurs during the study period.
Arm/Group | Simethicone Premedication | Placebo
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/27
Other Adverse Events (participants affected / at risk) | 0/27 | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No